CLINICAL TRIAL: NCT03661814
Title: Prophylactic Negative Pressure Wound Therapy to Reduce Surgical Site Infections in Elective Clean-Contaminated Colon Resections
Brief Title: Prophylactic NPWT to Reduce SSI in Colorectal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Kinetic Concepts, Inc. (Industry)
Responsible Party: Principal Investigator, joel bauer, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 18-0703
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Surgical Wound Infection
Keywords: Negative Pressure Wound Therapy; Colorectal Surgery; Prevena; Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Two cohorts. Experimental group receives the study device and the control group receives the standard of care (No device). Patients are randomized to either group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Prevena (Experimental): This group will receive the negative pressure wound therapy device.
  Interventions: Device: Prevena
- Standard of Care (No Intervention): This group will not receive the device and their surgery and clinical course will proceed as if they were not part of the study. They will receive the standard of care wound dressings.

INTERVENTIONS:
Device: Prevena — The NPWT device is a wound dressing with a vacuum system that can be placed over abdominal wounds, placed in the immediate postoperative period over abdominal wounds after clean/contaminated colorectal surgical procedures.
  Other Names: Negative pressure wound therapy device
  Arms: Prevena

SUMMARY:
The purpose of this study is to see if the Negative Pressure Wound Therapy (NPWT) system is effective and safe for the prevention of superficial and deep incisional surgical site infections (SSI) in high risk patients within 30 days after elective colorectal surgery. It has been shown that patients with an IBD, patients undergoing a reoperation or patients with certain comorbidities are at a higher risk of developing an SSI. The NPWT device is a wound dressing with a vacuum system that can be placed over abdominal wounds. The study will include up to 400 patients at this single site, where these high risk patients will be randomized to receive either one of two arms. The first arm involves the placement of the NPWT device in the immediate postoperative period over abdominal wounds after clean/contaminated colorectal surgical procedures. The device would then be left on for 5 days. The second arm would be standard of care and would entail routine postoperative protocols. Subjects will then be seen once at a 30 day (± 7 days) follow-up visit to assess for the development of SSIs.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-80
* patients who will undergo an open or laparoscopic-assisted clean/contaminated colorectal surgical procedure.
* Patients must either have an inflammatory bowel disease, undergoing reoperation within 30 days, or have two or more of the following risk factors: presence of an ostomy, type II diabetes, BMI greater than 30, immunosuppression, malnutrition, current smoker, chronic kidney disease (creatinine > 1.2), and disseminated cancer.

Exclusion Criteria:

* patients currently enrolled in another interventional clinical trial,
* patients with a BMI less than 20, patients with a current abdominal abscess or infection (including a known urinary tract infection),
* patients allergic to or hypersensitive to silver, patients planning to undergo a second colorectal surgical procedure (e.g., colostomy or ileostomy takedown) or any other general surgery in less than 30 days of index-surgery,
* any patient in which the planned surgery would include: i) placement of a stoma in the principal incision; ii) placement of a drain into the supra-peritoneal fascia space that emerges through the principal incision; iv) placement of a drain into the intraperitoneal space that emerges through the principal incision; and v) supplementation of any of the irrigation fluid with antibiotic or antiseptic drugs,
* patients with healing disorders,
* pregnant women,
* prisoners, or
* any patient that is deemed unsuitable for the study by the Principal Investigator or the operating surgeon/Co-Investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Bauer, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fry DE. The prevention of surgical site infection in elective colon surgery. Scientifica (Cairo). 2013;2013:896297. doi: 10.1155/2013/896297. Epub 2013 Dec 19. PMID 24455434
- [Background] Shepard J, Ward W, Milstone A, Carlson T, Frederick J, Hadhazy E, Perl T. Financial impact of surgical site infections on hospitals: the hospital management perspective. JAMA Surg. 2013 Oct;148(10):907-14. doi: 10.1001/jamasurg.2013.2246. PMID 23965750
- [Background] Tanner J, Padley W, Assadian O, Leaper D, Kiernan M, Edmiston C. Do surgical care bundles reduce the risk of surgical site infections in patients undergoing colorectal surgery? A systematic review and cohort meta-analysis of 8,515 patients. Surgery. 2015 Jul;158(1):66-77. doi: 10.1016/j.surg.2015.03.009. Epub 2015 Apr 25. PMID 25920911
- [Background] Bonds AM, Novick TK, Dietert JB, Araghizadeh FY, Olson CH. Incisional negative pressure wound therapy significantly reduces surgical site infection in open colorectal surgery. Dis Colon Rectum. 2013 Dec;56(12):1403-8. doi: 10.1097/DCR.0b013e3182a39959. PMID 24201395
- [Background] Chadi SA, Vogt KN, Knowles S, Murphy PB, Van Koughnett JA, Brackstone M, Ott MC. Negative pressure wound therapy use to decrease surgical nosocomial events in colorectal resections (NEPTUNE): study protocol for a randomized controlled trial. Trials. 2015 Jul 30;16:322. doi: 10.1186/s13063-015-0817-8. PMID 26223227

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from August 2018 - December 2018
Groups:
- Prevena: Prevena: The negative pressure wound therapy (NPWT) device is a wound dressing with a vacuum system that can be placed over abdominal wounds, placed in the immediate postoperative period over abdominal wounds after clean/contaminated colorectal surgical procedures.
Period: Overall Study
Arm/Group | Prevena | Standard of Care
Started | 2 | 5
Completed | 2 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prevena | Standard of Care | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (13.44) | 68.4 (8.38) | 64.7 (9.996)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Surgical Site Infection
Description: Any type of Surgical site infection as defined by the CDC developed within the follow-up period.
Time Frame: 37 days
Measure: Number; unit: incidences
Arm/Group | Prevena | Standard of Care
Number analyzed (Participants) | 2 | 5
incidences | 2 | 4

2. Secondary Outcome: Length of Hospital Stay
Time Frame: average of 7 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prevena | Standard of Care
Number analyzed (Participants) | 2 | 5
days | 7 (1.00) | 7.8 (2.71)

3. Secondary Outcome: Number of Serious Adverse Events
Description: Number of serious adverse events developed within the follow-up period
Time Frame: up to 37 days
Measure: Number; unit: events
Arm/Group | Prevena | Standard of Care
Number analyzed (Participants) | 2 | 5
events | 0 | 0

ADVERSE EVENTS:
Time Frame: 37 days
Arm/Group | Prevena | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 0/2 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03661814/Prot_SAP_000.pdf